CLINICAL TRIAL: NCT01396993
Title: Prospective Trial Evaluating Cosmetic And Oncologic Outcome Of Immediate Techniques For Oncoplastic Surgery In Breast Cancer
Brief Title: Prospective Non-randomized Evaluation of Oncoplastic Surgery
Acronym: iTOP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Florian Fitzal, Professor of Surgery, Medical University of Vienna
Other Study IDs: iTOP
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Breast Image Scale Index for Self Esteem Evaluation; Breast Symmetry Index; Quality of Life; Morbidity; Oncological Outcome
MeSH Terms: interventions — Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- iTOP: Patients undergoing immediate techniques for oncoplastic surgery (level I only parenchmyl rotation and breast undermining as well as level II using complex reduction plastics for nipple-areola-complex movings) and patients with mastectomy and immediate reconstruction
  Interventions: Procedure: Breast Surgery
- BCT: patients undergoing conservative breast surgery
  Interventions: Procedure: Breast Surgery

INTERVENTIONS:
Procedure: Breast Surgery — breast conserving surgery AND immediate defect filling using local flaps (level I) or reduction plastics (level II) as well as mastectomy and immediate reconstruction using free flaps
  Groups: iTOP
Procedure: Breast Surgery — Breast conserving therapy without defect correction
  Groups: BCT

SUMMARY:
Breast conserving therapy (BCT) is the standard treatment for intraductal or invasive breast cancer patients. However cosmetic results, e.g. symmetry and nipple displacement, are sometimes poor reducing the quality of life. The use of immediate techniques for oncoplastic surgery (iTOP) seems to improve subjective cosmetic outcome. Oncologic safety of iTOP has been demonstrated by several authors using restrospective analyses. However, no prospective observational trial has been done to objectively evaluate cosmetic and oncologic outcome comparing BCT with iTOP. The aim of this study is to investigate this issue within a prospective non randomized observational trial at the Medical University Vienna.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for unilateral breast conserving surgery due to cancer or a suspicious lesion, in whom >10%* of breast volume (measured by mammograms using a defined formular 37) has to be removed or breast cancer patients scheduled for mastectomy and immediate reconstruction (immediate or delayed contralateral correction is allowed)
* BIRADS IV, V or VI are eligible
* > 18 years of age
* Psychological and physical capable of understanding and performing the trial
* Signed written informed consent * If oncologic safety necessitates to resect more than half of one breast quadrant

Exclusion Criteria:

* Inflammatory breast cancer
* Progression after neoadjuvant therapy
* Pregnant women
* Patients unable to perform surgery under general anaesthesia
* Bilateral breast lesions

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a BIRADS IV, V or VI breast lesion are preoperatively asked to take part in this study if more than 10% of breast tissue will be excised or mastectomy and immediate reconstruction is planned. Patients with planned mastectomy without immediate reconstruction are not included. Patients scheduled for breast conservation can decide whether they undergo regular breast conservation (BCT) or BCT using immediate techniques of oncoplastic surgery (iTOP). A contralateral correction may be performed in both groups at any time of the trial. The use of a contralateral correction of patients without an immediate oncoplastic procedure does not initiate a change into the other group (intention to treat analyses).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-07 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
breast image scale | 2 years
  self esteem measured by the breast image scale will be assessed before and every 6 months after surgery as primary endpoint.

SECONDARY OUTCOMES:
quality of life | 2 years
  BREAST Q, non-validated questionnaires
Morbidity | 6 months
  Necrosis, infection, reoperations and bleedings as well as heamtoma and seroma formation will be clinically assessed after surgery
breast symmetry index | 2 years
  Using the breast analyzing tool software we will analyze breast symmetry before and every 6 months after surgery
oncologic parameters | 2-5 years
  local, distent and overal survival 2 as well as 5 years after surgery will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Austria